CLINICAL TRIAL: NCT03262727
Title: The Effect of BMS-986165 on the Pharmacokinetics of a Combined Oral Contraceptive (Ethinyl Estradiol/Norethindrone) in Healthy Female Subjects
Brief Title: The Effect of BMS-986165 Combined With an Oral Contraceptive (Ethinyl Estradiol/Norethindrone) in Healthy Female Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM011-039
Record Dates: First submitted 2017-08-24; First posted 2017-08-25 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Systemic Lupus Erythematosus; Arthritic Psoriasis; Psoriasis; Inflammatory Bowel Diseases
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis, Psoriatic; Psoriasis; Inflammatory Bowel Diseases | interventions — deucravacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BMS-986165 and Oral Contraceptive (Experimental): Oral administration of contraceptive, then progress to combination
  Interventions: Drug: BMS-986165; Drug: Loestrin 1.5/30 (1.5 mg norethindrone acetate/30 μg ethinyl estradiol)

INTERVENTIONS:
Drug: BMS-986165 — Oral administration of specified dose on specified days
Drug: Loestrin 1.5/30 (1.5 mg norethindrone acetate/30 μg ethinyl estradiol) — Oral Contraceptive

SUMMARY:
The purpose of this study is to investigate the effect of BMS-986165 in combination with an oral contraceptive in healthy female patients.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.0 and 32.0 kg/m2 inclusive,
* Weight ≥ 50 kg
* Negative result for tuberculosis (TB) as evidenced by a QuantiFERON-TB Gold Plus test at screening, or documentation of a negative result within 4 weeks before Cycle 1, Day 1
* Women of childbearing potential with intact ovarian function, on a stable regimen of combination birth control containing EE without evidence of clinically significant breakthrough bleeding or spotting for at least 2 consecutive months prior to Cycle 1 Day -1
* Subjects aged 21 years or older must have a normal Pap smear result within 3 years before Cycle 1 Day 1 (a Pap smear may be performed at screening if no result is available); a finding of abnormal squamous cells of unknown significance (ASCUS) is allowed provided it is an initial finding and not a follow up from an initial finding of ASCUS

Exclusion Criteria:

* Exposure to an investigational agent within 12 weeks before Cycle 1 Day 1
* Subjects who are pregnant or breastfeeding
* Any significant acute or chronic medical illness including infection, any active infection, febrile illness within 7 days before Cycle 1, Day 1, or any condition that could predispose the subject to infection
* History of recurrent or chronic sinusitis, bronchitis, pneumonia, urinary tract infection (recurrent or chronic urinary tract infection is 2 episodes within 6 months)
* Any serious acute or chronic bacterial, fungal, or viral infection (eg, pneumonia, septicemia) within the 3 months prior to screening
* Known or suspected autoimmune disorder, or any history of known or suspected congenital or acquired immunodeficiency state or condition that would compromise the subject's immune status (eg, history of splenectomy, primary immunodeficiency, etc)

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-11-23 (Actual); Study Completion 2017-12-19 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) derived from plasma concentration versus time | Approximately 1 day
Area under the plasma concentration-time curve to the end of the dosing period [AUC(tau)] derived from plasma concentration versus time | Approximately 1 day

SECONDARY OUTCOMES:
Adverse events measured by incidence | Approximately 86 days
Serious adverse events measured by incidence | Approximately 86 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Miami Research Associates, Miami, Florida, United States

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx